CLINICAL TRIAL: NCT00005978
Title: Dose Escalation Study of 131 I-Metaiodobenzylguanidine (MIBG) With Intensive Chemotherapy and Autologous Stem Cell Rescue for High-Risk Neuroblastoma - A Phase I Study
Brief Title: N99-01: Combination Chemotherapy, Radiation Therapy, and Stem Cell Transplantation in Treating Patients With Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Approaches to Neuroblastoma Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Katherine Matthay, MD, UCSF
Purpose: Treatment
Other Study IDs: CDR0000067966; P01CA081403 (NIH); N99-01 (Other: NANT Consortium)
Record Dates: First submitted 2000-07-05; First posted 2003-12-23 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2009-05

CONDITIONS: Neuroblastoma
Keywords: localized resectable neuroblastoma; regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; recurrent neuroblastoma; localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; Carboplatin; Etoposide; Melphalan; Peripheral Blood Stem Cell Transplantation; 3-Iodobenzylguanidine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: etoposide
Drug: melphalan
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: iobenguane I 131
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Giving the drugs in different ways may kill more tumor cells. Radiation therapy uses high-energy x-rays to damage tumor cells. Peripheral stem cell or bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy.

PURPOSE: This phase I trial is studying the side effects and best dose of combination chemotherapy when given before stem cell transplant and radiation therapy in treating patients with neuroblastoma that has not responded to previous treatments.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and toxic effects of iodine I 131 metaiodobenzylguanidine (131 I-MIBG) plus ablative doses of carboplatin and etoposide administered with fixed-dose melphalan followed by autologous hematopoietic stem cell transplantation in patients with refractory or residual high-risk neuroblastoma.
* Determine the number of days until blood counts recover in these patients after receiving this treatment regimen.
* Determine the response rate to this treatment regimen in these patients.
* Determine the tumor dosimetry of 131 I-MIBG in patients with measurable soft tissue lesions.

OUTLINE: This is a dose-escalation study of iodine I 131 metaiodobenzylguanidine (131 I-MIBG), carboplatin, and etoposide. Patients are stratified according to glomerular filtration rate (at least 100 mL/min vs 60-99 mL/min).

Patients undergo peripheral blood stem cell harvest or bone marrow harvest at least 2 weeks prior to treatment with 131 I-MIBG.

Patients receive 131 I-MIBG IV over 120 minutes on day -21; melphalan IV on days -7 to -5; carboplatin and etoposide IV continuously over 96 hours on days -7 to -4; autologous hematopoietic stem cell transplantation IV over 15-30 minutes on day 0; and filgrastim (G-CSF) subcutaneously or IV starting on day 0 and continuing until blood counts recover. Radiotherapy is administered to the primary tumor site and metastatic sites twice daily for 7 consecutive days within 6 weeks of transplantation or once blood counts have recovered.

Cohorts of 3-6 patients receive escalating doses of 131 I-MIBG, carboplatin, and etoposide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at day 84, and then 2 months later if there is a complete response and/or partial response. Patients who continue therapy on other protocols are followed before starting the new therapy. All patients are followed for life for any delayed toxic effects related to study therapy, secondary malignancies, disease status, and survival.

PROJECTED ACCRUAL: A total of 30-60 patients (15-30 per stratum) will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neuroblastoma as evidenced by one of the following:

  * Histological confirmation
  * Demonstrates clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites
* High-risk refractory or residual disease
* Poorly responding disease, meeting 1 of the following criteria:

  * Stable disease or partial response after at least 12 weeks of induction therapy
  * Bone marrow containing greater than 100 tumor cells per 100,000 normal cells after 12 weeks of induction therapy
  * Progressive disease during or after therapy
* At least 1 prior positive iodine I 131 metaiodobenzylguanidine (131 I-MIBG) scan since diagnosis and meets disease status criteria

PATIENT CHARACTERISTICS:

Age:

* 1 to 21 (1 to 20 at diagnosis)

Performance status:

* ECOG 0-2

Life expectancy:

* At least 2 months

Hematopoietic:

* Absolute neutrophil count at least 500/mm^3
* Platelet count at least 20,000/mm^3 (transfusion allowed)
* Hemoglobin at least 8 g/dL (transfusion allowed)

Hepatic:

* Bilirubin normal
* AST/ALT no greater than 3 times normal
* No active hepatitis (for HIV-positive patients only)

Renal:

* Glomerular filtration rate or creatinine clearance at least 60 mL/min
* Creatinine less than 1.5 times normal for age

Cardiovascular:

* Ejection fraction at least 55% OR
* Fractional shortening at least 30%

Pulmonary:

* No dyspnea at rest or exercise intolerance
* No requirement for supplemental oxygen
* No active pneumonia (for HIV-positive patients only)

Other:

* No disease of any major organ system that would preclude study participation
* No other active health problems (for HIV-positive patients only)
* No active infections requiring intravenous antivirals, antibiotics, or antifungals
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic therapy and recovered

Chemotherapy:

* At least 3 weeks since prior chemotherapy and recovered
* No more than 100 mg/m^2 total dose of prior melphalan

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior total body, whole abdominal, or whole liver irradiation
* No prior therapy with 131 I-MIBG
* At least 2 weeks since prior radiotherapy (6 months for prior radiotherapy to craniospinal or whole lung fields or greater than 50% of bone marrow space) and recovered

Surgery:

* Prior surgical resection allowed
* Recovered from prior surgery

Other:

* No prior myeloablative therapy

  * Prior submyeloablative therapy with peripheral blood stem cell support allowed
* No concurrent antiretrovirals for HIV-positive patients
* Concurrent prolonged antifungal allowed if culture and biopsy negative in suspected residual radiographic lesions
* No medications that may preclude uptake of 131 I-MIBG for 1 week prior and 2 weeks after administration of study drugs
* No concurrent hemodialysis

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2000-05; Primary Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine K. Matthay, MD, Study Chair — Children's Hospital Los Angeles
Locations (15):
- United States (15):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Cancer Center, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Matthay KK, Tan JC, Villablanca JG, Yanik GA, Veatch J, Franc B, Twomey E, Horn B, Reynolds CP, Groshen S, Seeger RC, Maris JM. Phase I dose escalation of iodine-131-metaiodobenzylguanidine with myeloablative chemotherapy and autologous stem-cell transplantation in refractory neuroblastoma: a new approaches to Neuroblastoma Therapy Consortium Study. J Clin Oncol. 2006 Jan 20;24(3):500-6. doi: 10.1200/JCO.2005.03.6400. PMID 16421427